CLINICAL TRIAL: NCT03509233
Title: Anti-infectious Therapy of Chronic Periodontitis Using One Stage Full Mouth Disinfection With Subgingival Airpolishing - a Comparison of Different Clinical Strategies
Brief Title: Anti-infectious Therapy of Periodontitis - Comparison of Different Clinical Strategies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Principal Investigator, Sareh Michael, Dr. med., RWTH Aachen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RWTHAachenUParo01
Record Dates: First submitted 2018-03-20; First posted 2018-04-26 (Actual); Last update posted 2020-08-31 (Actual); Status verified 2020-08

CONDITIONS: Periodontitis
Keywords: periodontitis; full mouth scaling; air abrasion; scaling
MeSH Terms: conditions — Periodontitis | interventions — N(3)-(4-methoxyfumaroyl)-2,3-diaminopropionic acid

STUDY DESIGN:
Intervention Model Description: multicenter randomized controlled intervention trial
Who Masked: Investigator
Masking Description: The examiner performing the measurement of all clinical periodontal parameters is not aware of the type of treatment provided to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Q-SRP (Active Comparator): Quadrant scaling and root planing
  Interventions: Other: Q-SRP
- FMS (Experimental): Full mouth scaling and root planing
  Interventions: Other: FMS
- FMD (Experimental): Full mouth disinfection
  Interventions: Other: FMD
- FMDP (Experimental): Full mouth disinfection with periopolishing
  Interventions: Other: FMDP

INTERVENTIONS:
Other: Q-SRP — Quadrant scaling and root planing under local anesthesia using ultrasonic devices (Piezon-Master, EMS) and Gracey curettes (Hu-Friedy) within four sessions in intervals of 1 week
  Arms: Q-SRP
Other: FMS — Full mouth scaling and rootplaning under local anesthesia using ultrasonic devices (Piezon-Master, EMS) and Gracey curettes (Hu-Friedy) within 24 hours
  Arms: FMS
Other: FMD — Full mouth scaling and rootplaning under local anesthesia using ultrasonic devices (Piezon-Master, EMS) and Gracey curettes (Hu-Friedy) within 24 hours with additional disinfection using 0.2% chlorhexidine (mouth rinsing and tonsil spray), subgingival application of 1% chlorhexidine gel and 2 months postoperative home care using chlorhexidine 0.2% (rinse and spray)
  Arms: FMD
Other: FMDP — FMD protocol (see FMD arm) with additional use of subgingival airpolishing (Air Flow, EMS) using Erythritol powder (Air-Flow Plus powder, EMS) for 20 seconds per tooth
  Arms: FMDP

SUMMARY:
It is the aim of the study to evaluate the efficiency of "One stage full mouth disinfection" according to the original protocol (Quirynen et al. 1995) in comparison to other approaches considering different scaling strategies and different disinfection concepts. Therefore, a multicenter randomized control treatment will be performed. In total, 204 patients with chronic periodontitis shall be allocated to the following treatment concepts. Group A: quadrant scaling with weekly intervals (Q-SRP; N = 51); Group B: full mouth scaling (FMS; N = 51); Group C: full mouth disinfection (FMD; N = 51); Group D: full mouth disinfection with subgingival glycine air polishing using erythritol powder (FMDP; N = 51). Evaluation of periodontopathic parameters and periodontal pathogens at baseline, 3 months and 6 months shall give evidence about the benefits of concept and the single components of FMD.

ELIGIBILITY:
Inclusion Criteria:

* patients with generalized moderate to severe chronic periodontitis
* presence of at least 18 teeth
* with at least 2 multi-rooted and / or 2 single-rooted teeth in the first quadrant with at least 6 sites with periodontal probing depth of ≥ 6 mm
* radiographic bone loss of at least 25% of the root length

Exclusion Criteria:

* subgingival scaling and root planing within the last 12 months
* antimicrobial rinsing or intake of systemic antibiotics within the last 4 months
* systemic diseases with known interactions to periodontal disease or known need for antibiotic prophylaxis
* known intolerance / allergies to chlorhexidine
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03-27 (Actual); Study Completion 2020-08-27 (Actual)

PRIMARY OUTCOMES:
Change of clinical attachment level | Baseline, 3 months, 6 months
  Measuring the change of the distance between the cemento-enamel junction and the bottom of the periodontal pocket 3 and 6 months after therapy compared to baseline

SECONDARY OUTCOMES:
Change of pocket probing depth | Baseline, 3 months, 6 months
  Measuring the change of the distance between the gingival sulcus and the bottom of the periodontal pocket 3 and 6 months after therapy compared to baseline
Change of presence of periodontopathogenic bacteria A. actinomycetemcomitans, P. gingivalis, P. intermedia and T. denticola | Baseline, 3 months, 6 months
  Analysis of pooled subgingival plaque specimen for the presence of periodontopathogenic marker bacteria A. actinomycetemcomitans, P. gingivitis, T. forsythia and P. intermedia; Assessment of the change of the occurrence of these bacteria 3 and 6 months after therapy compared to baseline
Change of bleeding on probing | Baseline, 3 months, 6 months
  Assessment of the change of the appearance of a bleeding spot immediately after the probing of periodontal pockets 3 and 6 months after therapy compared to baseline
Change of gingival index | Baseline, 3 months, 6 months
  Recording the change of the presence of supragingival plaque according to the criteria by assessment of the inflammatory status of the gingiva according to Löe et al. 3 and 6 months after therapy compared to baseline
Change of plaque index | Baseline, 3 months, 6 months
  Recording the change of the presence of supragingival plaque according to the criteria by Silness and Loe 3 and 6 months after therapy compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Jamal M. Stein, Prof. Dr., Study Director — Universitätsklinikum RWTH Aachen
Locations (5):
- Germany (4):
  - Universitätsklinikum RWTH Aachen, Klinik für Zahnerhaltung, Parodontologie u. Präventive Zahnheilkunde, Aachen
  - Charité Centrum Zahn-, Mund- und Kieferheilkunde, Parodontologie und Synoptische Zahnmedizin, Berlin
  - Universitätspoliklinik für Zahnerhaltungskunde und Parodontologie, Halle
  - Universitätsmedizin Mainz, Poliklinik f. Zahnerhaltung u. Parodontologie, Mainz
- Department of Dental Medicine 1 (Periodontology), Timișoara, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdelbary MMH, Schittenhelm F, Yekta-Michael SS, Reichert S, Schulz S, Kasaj A, Braun A, Conrads G, Stein JM. Impact of Three Nonsurgical, Full-Mouth Periodontal Treatments on Total Bacterial Load and Selected Pathobionts. Antibiotics (Basel). 2022 May 19;11(5):686. doi: 10.3390/antibiotics11050686. PMID 35625330
- [Derived] Schulz S, Stein JM, Schumacher A, Kupietz D, Yekta-Michael SS, Schittenhelm F, Conrads G, Schaller HG, Reichert S. Nonsurgical Periodontal Treatment Options and Their Impact on Subgingival Microbiota. J Clin Med. 2022 Feb 23;11(5):1187. doi: 10.3390/jcm11051187. PMID 35268280
- [Derived] Stein JM, Yekta-Michael SS, Schittenhelm F, Reichert S, Kupietz D, Dommisch H, Kasaj A, Wied S, Vela OC, Stratul SI. Comparison of three full-mouth concepts for the non-surgical treatment of stage III and IV periodontitis: A randomized controlled trial. J Clin Periodontol. 2021 Dec;48(12):1516-1527. doi: 10.1111/jcpe.13548. Epub 2021 Oct 4. PMID 34517434